CLINICAL TRIAL: NCT00404391
Title: A Randomized, Double-Blind, Placebo-Controlled Study Comparing the Analgesic Activity of Hydrocodone/Acetaminophen Extended Release and Placebo in Subjects With Pain Following Bunionectomy Surgery
Brief Title: A Study Comparing the Analgesic Activity of Extended Release Hydrocodone/Acetaminophen (Vicodin® CR) and Placebo in Subjects With Pain Following Bunionectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Victor Jorden, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-609
Record Dates: First submitted 2006-11-26; First posted 2006-11-28 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pain
Keywords: Moderate to severe pain following bunionectomy surgery
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: Hydrocodone/Acetaminophen Extended Release
- Arm 2: hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: Hydrocodone/Acetaminophen Extended Release
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen Extended Release — 1 tablet every 12 hours
  Other Names: ABT-712
  Arms: Arm 1: hydrocodone/acetaminophen extended release
Drug: Hydrocodone/Acetaminophen Extended Release — 2 tablets every 12 hours
  Other Names: ABT-712
  Arms: Arm 2: hydrocodone/acetaminophen extended release
Drug: Placebo — 2 tablets every 12 hours
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of the administration of 2 different dose levels of Extended Release Hydrocodone/Acetaminophen with placebo over a 48 hour dosing period in patients who have had bunionectomy surgery, and to assess the safety of the drug for 7 days after patients are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 to 65
* Females must be of non-childbearing potential or practicing birth control
* Subject is scheduled to undergo primary, unilateral first metatarsal bunionectomy surgery

Exclusion Criteria:

* Is allergic to or has a serious reaction to hydrocodone, or other opioids, acetaminophen, lidocaine or propofol, and/or similar drugs
* Has initiated corticosteroid therapy within the past month or is scheduled to receive any corticosteroid during the study
* Is associated with any currently ongoing research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2003-10; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Time-interval-weighted sum of pain relief (TOTPAR)score for 0 to 12 hours following the first dose of study drug administration | 12 hours
  Pain relief measured by a 100mm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Time interval weighted sum of pain intensity difference (SPID)scores | 12 hours
  Sum of pain intensity difference

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — Abbott
Locations (4):
- United States (4):
  - Site Ref # / Investigator 4993, Owing Mills, Maryland
  - Site Ref # / Investigator 4994, Austin, Texas
  - Site Ref # / Investigator 4992, San Marcos, Texas
  - Site Ref # / Investigator 4995, Salt Lake City, Utah